CLINICAL TRIAL: NCT04688697
Title: A Multicentric, Open-labeled, Prospective, Randomized Controlled Study to Compare the Satisfaction and Safety of the Prepectoral and Subpectoral Implant-based Breast Reconstruction in Patients Receiving Immediate Breast Reconstruction Using Implant Combined With TiLoop® Bra After Skin Sparing or Nipple-areola Sparing Mastectomy
Brief Title: Prepectoral and Subpectoral Implant-based Breast Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiong Wu, Professor, Vise President, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIBBR
Record Dates: First submitted 2020-12-25; First posted 2020-12-30 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Breast Carcinoma; Breast Reconstruction
Keywords: breast carcinoma; breast reconstruction; Prepectoral prosthetic breast reconstruction; Complication
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prepectoral Group (Experimental): Prepectoral implant-based reconstruction applied for patients in this group
  Interventions: Procedure: prepectoral implant-based reconstruction
- Subpectoral Group (Active Comparator): Subpectoral implant-based reconstruction applied for patients in this group
  Interventions: Procedure: subpectoral implant-based reconstruction

INTERVENTIONS:
Procedure: prepectoral implant-based reconstruction — In this group, patients receive breast reconstruction with prosthesis placed to anterior pectoralis major, synthetic mesh is used to enclose the prosthesis and place it to anterior pectoralis major.
  Arms: Prepectoral Group
Procedure: subpectoral implant-based reconstruction — In this group, patients receive breast reconstruction with placed to posterior pectoralis major, part of the mesh is placed under the pectoralis major during the operation, and the mesh is used to cover the suture of the prosthesis on the inferior plica, or to directly enclose the lower part of the implant.
  Arms: Subpectoral Group

SUMMARY:
Breast cancer is one of the main malignant tumors threatening women's lives. In recent years, the increasing demand for reconstruction of breast cancer patients in China has made the proportion of breast reconstruction increase year by year, while implant reconstruction has become the most important way of breast reconstruction due to its less injury, shorter time of operation and relatively simple surgical technique. In the long-term clinical practice, due to the lack of safe and effective alternative methods, the reconstruction method with prosthesis placed to posterior pectoralis major has been accepted by surgeons and patients, and has become the most commonly used method of prosthesis construction. However, the development of biomaterials provides new ideas for breast reconstruction. At present, more and more doctors in clinical practice discontinue the use of serratus anterior, but use the synthetic mesh (mostly titanium mesh TiLoop® Bra) or allogeneic acellular dermal matrix mesh to cover part of the dilator or prosthesis so as to shorten the entire operation cycle and make the appearance of the reconstructed breast more natural and aesthetic. In particular, it can improve the contour of the folds under the breast and shape the breasts with a certain degree of sagging.

This study takes the patients receiving immediate reconstruction with an implant combined with TiLoop® Bra after total mastectomy as the subjects, aiming to compare the aesthetics and safety of the placement of implant to anterior and posterior pectoralis major through a prospective and randomized study. The primary objective of the study is to analyze the aesthetics of breast appearance, patient satisfaction and postoperative quality of life (QOL) of the placement of implant to anterior and posterior pectoralis major. The secondary objective of the study is to analyze the incidence of complications and type of reoperation in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years old
2. Female
3. Preoperative pathology confirming invasive breast carcinoma or ductal carcinoma in situ
4. Clinical T1 and T2 (Maximum tumor diameter ≤5 cm)
5. Clinical ALN negative (Clinical physical examination and ultrasound indicate axillary lymph node negative; Suspected abnormality of axillary lymph node, and fine needle aspiration negative)
6. No clinical or imaging evidence of distant metastasis
7. Patients to receive skin sparing mastectomy or nipple sparing mastectomy
8. BMI < 35
9. Patients with no or mild mastoptosis
10. Prosthesis to be implanted <500 ml
11. Be able and willing to sign the Informed Consent Form (ICF)

Exclusion Criteria:

1. Patients with the breast of moderate-severe mastoptosis, or requiring the use of Wise-pattern or other breast lift methods for subcutaneous mammary gland resection
2. BMI>=35
3. Patients who have received symmetrical breast surgery on the unaffected side immediately or later
4. Patients with locally advanced breast cancer to receive neoadjuvant therapy
5. Patients currently participating in other clinical trials, which may have impact on the participation in this trial
6. Neoadjuvant therapy has been completed, and there is clear indication of adjuvant radiotherapy after the operation
7. Previous history of breast cancer (patients with ipsilateral recurrence after breast sparing surgery)
8. Pregnancy breast-feeding women
9. History of smoking
10. Previous history of diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients' satisfaction | 18 months after the operation
  Patients' satisfaction evaluated based on Breast-Q scale

SECONDARY OUTCOMES:
Incidences of complications and serious complications | During 18 months after the operation
  Incidences of complications and serious complications

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided